CLINICAL TRIAL: NCT04542434
Title: A Phase 2 Randomized Double Blind, Placebo-controlled Study on the Safety and Efficacy of Niclosamide in Patients With COVID-19
Brief Title: Niclosamide in COVID-19
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor asset acquired by another pharma company who opened their own IND for this compound. First Wave Bio never started this study in the US or ex-US.
Sponsor: Entero Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FW-COV-003
Record Dates: First submitted 2020-09-04; First posted 2020-09-09 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2021-12

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Niclosamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Niclosamide (Experimental)
  Interventions: Drug: Niclosamide Oral Tablet
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Niclosamide Oral Tablet — Niclosamide tablets 400 mg 3 times daily for 14 days
  Arms: Niclosamide
Drug: Placebo — Matching placebo tablets 3 times daily for 14 days
  Arms: Placebo

SUMMARY:
This is a two-part, Phase 2, multicentre, randomized, double blind, 2-arm placebo-controlled study in adults with moderate COVID-19 with gastrointestinal signs and symptoms

ELIGIBILITY:
Inclusion Criteria:

* Part 1 only: Patients hospitalized with a primary diagnosis of COVID-19 with or without pneumonia, who are expected to remain in hospital at least seven days after the randomization and who accept continuing to be assessed for the study procedures (home or outpatient unit) up to 6 weeks in case of discharge.

Part 2 only: Patients with a primary diagnosis of COVID-19 with or without pneumonia who are not planned to be hospitalized.

* Patients who prior to developing COVID-19 usually have normal bowel habits defined as at least solid-formed 3 stools per week and no more than 3 solid-formed stools per day.
* SARS-CoV-2 RNA presence in rectal swab (or stool test) ≤2 days before randomization by local or central lab.
* Diarrhea defined as at least 3 watery stools in the last 24 hours prior to enrolment

Exclusion Criteria:

* At the time of randomization patients requiring ICU admission or patients with severe respiratory insufficiency requiring mechanical ventilation or with rapid worsening of respiratory function leading to expectation for mechanical ventilation or ICU admission.
* Evidence of rapid clinical deterioration or existence of any life-threatening co-morbidity or any other medical condition which, in the opinion of the investigator, makes the patient unsuitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Mortality | From Day 1 to 6 weeks
  All-cause mortality
TEAE | From Day 1 to 6 weeks
  Proportion of patients with Treatment Emergent Adverse Events (TEAE) leading to study drug discontinuation
SAEs | From Day 1 to end of study
  Serious adverse event (SAE) coded by System Organ Class (SOC) and Preferred Term (PT), using the Medical Dictionary for Regulatory Activities (MedDRA)
Safety laboratory | From Day 1 to 6 weeks
  Change in safety laboratory tests from baseline to 6 weeks, the number of subjects with values low, normal, and high compared to the normal ranges pretreatment versus post-treatment will be provided
Blood pressure | From Day 1 to 6 weeks
  Change in sitting systolic and diastolic blood pressure from baseline to 6 weeks summarized descriptively by visit and presented as shift tables
fecal RNA virus clearance | From Day 1 to 6 weeks
  time to fecal RNA virus clearance (rectal swab or stool sample) assessed by RT-qPCR in the niclosamide group, compared to the placebo group (Part 2 only)
Body temperature | From Day 1 to 6 weeks
  Change in body temperature from baseline to 6 weeks summarized descriptively by visit and presented as shift tables
Heart rate | From Day 1 to 6 weeks
  Change in heart rate from baseline to 6 weeks summarized descriptively by visit and presented as shift tables
SaO2 | From Day 1 to 6 weeks
  Change in SaO2 from baseline to 6 weeks summarized descriptively by visit and presented as shift tables
ECG | From Day 1 to 6 weeks
  Change in ECG parameters including: 1. PR interval 2. RR interval 3. QRS interval 4 QT interval 5. HR interval 6. QtcF interval. All intervals summarized descriptively by visit from baseline to 6 weeks